CLINICAL TRIAL: NCT02484092
Title: Gene Therapy, Open-label, Dose-escalation Study of PF-06838435 (SPK-9001) [Adeno-associated Viral Vector With Human Factor IX Gene] in Subjects With Hemophilia B
Brief Title: A Gene Therapy Study for Hemophilia B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C0371005; SPK-9001-101 (Other: Alias Study Number)
Record Dates: First submitted 2015-06-18; First posted 2015-06-29 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; Blood Coagulation Disorders; Gene Therapy; Gene Transfer; Factor IX Deficiency; Factor IX Gene; Factor IX Protein; Vector; AAV
MeSH Terms: conditions — Hemophilia B; Blood Coagulation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPK-9001 (Experimental): Single intravenous (i.v.) infusion of SPK-9001 [an adeno-associated viral (AAV) vector with human factor IX gene] Intervention: Gene Therapy / Gene Transfer
  Interventions: Biological: SPK-9001

INTERVENTIONS:
Biological: SPK-9001 — A novel, bioengineered adeno-associated viral vector carrying human factor IX variant

SUMMARY:
A Phase 1/2, Open-Label, Non-Randomized, Dose-Escalation Study of SPK-9001 in Subjects with Hemophilia B.

DETAILED DESCRIPTION:
Hemophilia B, or Christmas disease, is a genetic bleeding disorder resulting in the lack of ability to produce blood-clotting factor IX (FIX). Individuals with hemophilia B suffer repeated bleeding events, which can cause chronic joint disease and sometimes leads to death due to the inability for blood to clot efficiently. This chronic joint disease can have significant physical, psychosocial, and quality-of-life effects, including financial burden. The current treatment is intravenous infusion of FIX protein products, either prophylactically or in response to bleeding.

The approach being tested in this study uses a novel recombinant adeno-associated virus (AAV), which in nature causes no disease, to deliver the human factor IX (hFIX) gene to the liver cells where FIX is normally made. Recent data of a gene therapy study showed preliminary encouraging results with the approach of using an AAV vector carrying the factor IX gene. This study will seek to determine the safety and kinetics of a single IV infusion of SPK-9001 (a novel AAV vector carrying a high specific activity factor IX variant).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent and comply with requirements of the study
* Males ≥18 y.o. with confirmed diagnosis of hemophilia B (≤2 IU/dL or ≤2% endogenous factor IX)
* Received ≥50 exposure days to factor IX products
* A minimum average of 4 bleeding events per year requiring episodic treatment of factor IX infusions or prophylactic factor IX infusions
* No measurable factor IX inhibitor as assessed by the central laboratory and have no prior history of inhibitors to factor IX protein
* Agree to use reliable barrier contraception until 3 consecutive samples are negative for vector sequences

Exclusion Criteria:

* Evidence of active hepatitis B or C
* Currently on antiviral therapy for hepatitis B or C
* Have significant underlying liver disease
* Have serological evidence* of HIV-1 or HIV-2 with CD4 counts ≤200/mm3 (* subjects who are HIV+ and stable with CD4 count >200/mm3 and undetectable viral load are eligible to enroll)
* Neutralizing antibodies reactive with AAV-Spark100 above and/or below a defined titre
* Participated in a gene transfer trial within the last 52 weeks or in a clinical trial with an investigational drug within the last 12 weeks
* Unable or unwilling to comply with study assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Genetic Males
Enrollment: 15 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (9):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC Davis CTSC Clinical Research Center, Sacramento, California
  - UC Davis Ellison Ambulatory Care Clinic, Sacramento, California
  - UC Davis Investigational Pharmacy, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Royal Prince Alfred Hospital, Camperdown/Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Pittman DD, Carrieri C, Soares H, McKay J, Tan CY, Liang JZ, Rakhe S, Marshall JC, Murphy JE, Gaitonde P, Rupon J. Field Study and Correlative Studies of Factor IX Variant FIX-R338L in Participants Treated with Fidanacogene Elaparvovec. Thromb Haemost. 2024 Oct;124(10):912-921. doi: 10.1055/s-0044-1787734. Epub 2024 Jun 11. PMID 38863155
- [Derived] George LA, Sullivan SK, Giermasz A, Rasko JEJ, Samelson-Jones BJ, Ducore J, Cuker A, Sullivan LM, Majumdar S, Teitel J, McGuinn CE, Ragni MV, Luk AY, Hui D, Wright JF, Chen Y, Liu Y, Wachtel K, Winters A, Tiefenbacher S, Arruda VR, van der Loo JCM, Zelenaia O, Takefman D, Carr ME, Couto LB, Anguela XM, High KA. Hemophilia B Gene Therapy with a High-Specific-Activity Factor IX Variant. N Engl J Med. 2017 Dec 7;377(23):2215-2227. doi: 10.1056/NEJMoa1708538. PMID 29211678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 22 participants were screened, 15 participants were assigned to treatment and completed study. All 15 participants received the lowest dose in the study (5 x 10^11 vg/kg). No participants were assigned to the 2 higher dose arms. Results presented here are from the lowest dose level.
Groups:
- SPK-9001 (5 x 10^11 vg/kg) IV Infusion: Participants were infused with 100 IU/kg of their usual FIX protein product over 10 minutes at Day 0 visit. Following the bolus infusion of the usual FIX protein product, the participant was infused with SPK-9001 (5 x 10^11 vg/kg) for approximately 60 minutes via infusion pump.
Period: Overall Study
Arm/Group | SPK-9001 (5 x 10^11 vg/kg) IV Infusion
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Arm/Group | SPK-9001 (5 x 10^11 vg/kg) IV Infusion
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 12
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 1
  Multiple | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Findings
Description: Physical examination included examination of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination assessed the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Findings were considered to be clinically significant based on investigator's decision.
Time Frame: Baseline up to Week 52
Population: All participants who received the infusion of SPK-9001.
Measure: Count of Participants; unit: Participants
Groups:
- SPK-9001 (5 x 10^11 vg/kg): Participants were infused with 100 IU/kg of their usual FIX protein product over 10 minutes at Day 0 visit. Following the bolus infusion of the usual FIX protein product, the participant was infused with SPK-9001 (5 x 10^11 vg/kg) for approximately 60 minutes via infusion pump.
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Participants | 0

2. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs (temperature, respiratory rate, pulse rate, height, weight, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline up to Week 52
Population: All participants who received the infusion of SPK-9001.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Participants | 0

3. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAE
Description: Following parameters were analyzed for laboratory examination: hematology (neutrophils, lymphocytes, monocytes, eosinophils, basophils, red blood cell [RBC] count, hemoglobin, hematocrit, platelet count); liver function (albumin, total bilirubin, total protein, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, alkaline phosphatase, GGT); Lipid panel (HDL, VLDL, triglycerides, total cholesterol); clinical chemistry (sodium, potassium, chloride, bicarbonate, glucose, phosphate, serum creatinine, BUN); urinalysis (specific gravity, pH, glucose, protein, blood, ketones; coagulation, immunology, etc. Investigators determined which laboratory abnormalities were reported as treatment-emergent adverse events (TEAEs).
Time Frame: Baseline up to Week 52
Population: All participants who received the infusion of SPK-9001.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Participants | 2

4. Primary Outcome: Number of Participants With Drug -Related TEAEs and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and AEs. An AE was regarded as TEAE if the start date was on or after the infusion of SPK-9001 but before participant's last visit on study (or the date of withdrawal/the date of being lost to follow-up). Severe TEAEs were TEAEs that interfered significantly with participants' usual function. Treatment-related TEAEs were determined by the investigator.
Time Frame: Baseline up to Week 52
Population: All participants who received the infusion of SPK-9001.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Participants
  Drug-related TEAE | 2
  Drug-related Serious TEAE | 0

5. Primary Outcome: Number of Participants With Positive Immune Reponses Against Adeno-associated Virus Vector (AAV) Capsid
Description: Peripheral blood mononuclear cells (PBMC) results by interferon gamma enzyme-linked immunospot assay (ELISPOT) to assess cellular immune responses to AAV capsid and to FIX were presented. The ELISPOT is a type of assay that focuses on quantitatively measuring the frequency of cytokine secretion for a single cell. The positive ELISPOT results suggested a T-cell reaction to capsid protein.
Time Frame: Baseline up to Week 52
Population: All participants who received the infusion of SPK-9001.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Participants | 2

6. Primary Outcome: Number of Participants Who Reached > 150% Vector-derived FIX:C Activity Level After SPK-9001 Infusion
Description: Based on non-clinical studies in non-human primates (NHPs), it was not predicted that vector-derived FIX:C activity levels >150% of normal would be achieved in this study. However, thrombin antithrombin (TAT) levels as thrombotic potential were to be measured if vector derived FIX:C activity levels >150% of normal were achieved in any participant during the study. Blood samples for TAT at Day 0 visit (prior to FIX protein product infusion) were used to establish baseline value.
Time Frame: Baseline up to Week 52
Population: All participants who received the infusion of SPK-9001.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Participants | 0

7. Primary Outcome: Number of Participants With FIX Inhibitor
Description: FIX inhibitors were measured using the Bethesda assay from the central and local laboratory. The Bethesda assay measures the amount of factor (FIX) inactivated when the plasma from the patient is incubated with an external source of factor for 2 hours at 37ºC. Inhibitor levels are quantified in Bethesda units (BU). An inhibitor titer of ≥ 0.6 BU/ml is to be taken as clinically significant.
Time Frame: Baseline up to Week 52
Population: All participants who received the infusion of SPK-9001.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Participants | 0

8. Primary Outcome: Incremental Recovery of FIX Product
Description: Incremental recovery was determined as the peak factor level recorded within the first 3 hours after infusion and was reported as (IU/ml)/(IU/kg), using the formula:([Activity IU/mL peak post infusion] - [Activity IU/mL pre-infusion]) / (IU/kg infused).
Time Frame: Day 0 and Week 52
Population: Participants who had received 100 IU/kg of FIX protein product infusion and completed the blood sample collection within the first 3 hours post infusion for FIX protein product enabling determination of FIX incremental recovery.
Measure: Mean (Standard Deviation); unit: [IU/ml]/[IU/kg]
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
[IU/ml]/[IU/kg]
  Day 0 | 0.0100 (0.00242)
  Week 52: number analyzed (Participants) | 6
  Week 52 | 0.0162 (0.01351)

9. Secondary Outcome: FIX:C Activity
Description: All samples collected from participants for plasma FIX activity levels were analyzed and used to determine peak and steady-state vector-derived circulating FIX activity levels. The vector-derived endogenous (not affected by intercurrent FIX product infusions) FIX:C activity levels were characterized by post-treatment population mean. Dose escalation and dose level expansion strategies were employed in the study based on vector-derived FIX activity levels as well as any immune responses against AAV capsid. Steady-state levels were based on 2 separate vector-derived FIX:C activity level measurements (at least 2 weeks apart) starting from Week 8-12 with adequate washout.
Time Frame: Baseline up to Week 52
Population: Participants who had received SPK-9001 and had collected vector-derived FIX:C activity levels enabling acceptable determination of the peak and steady-state derived activity level.
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Percentage of Normal
  Steady-State Level | 22.9 (9.89)
  Peak Activity | 29.1 (11.63)

10. Secondary Outcome: Change From Baseline in FIX:C Antigen Level at Steady State
Description: The vector-derived endogenous (not affected by intercurrent FIX product infusions) FIX:C activity antigen levels were characterized by post-treatment population mean.
Time Frame: Week 12 up to Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | SPK-9001 (5 x 10^11 vg/kg)
Number analyzed (Participants) | 15
Percentage of Normal
  Week 12 | -4.4 (19.26)
  Week 14: number analyzed (Participants) | 14
  Week 14 | -4.7 (23.11)
  Week 16 | -4.7 (19.79)
  Week 18 | -5.8 (21.81)
  Week 22 | -4.6 (22.06)
  Week 26 | -6.6 (20.64)
  Week 32: number analyzed (Participants) | 14
  Week 32 | -7.1 (20.48)
  Week 42 | -4.9 (19.87)
  Week 52 | -6.9 (19.70)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Arm/Group | SPK-9001 (5 x 10^11 vg/kg) IV Infusion
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPK-9001 (5 x 10^11 vg/kg) IV Infusion (N=15)
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Food poisoning (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Catheter site bruise (General disorders) | 1
Face oedema (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Ligament sprain (Injury, poisoning and procedural complications) | 1
Muscle injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 3
Transaminases increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Calcification of muscle (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
15 participants were treated at the first dose planned for this dose escalation study. Requirements for dose escalation were not met as per protocol and the study completed once all participants completed 52 weeks of follow-up at the initial dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT02484092/SAP_000.pdf
  • Study Protocol (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT02484092/Prot_001.pdf